CLINICAL TRIAL: NCT01663948
Title: International Plastic Bronchitis Registry
Status: Terminated | Type: Observational
Why Stopped: Loss of staff combined with low study enrollment and a change in lab/PI priorities
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM14554
Record Dates: First submitted 2012-08-09; First posted 2012-08-14 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Plastic Bronchitis
Keywords: Plastic bronchitis; PB

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Airway Casts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Plastic bronchitis

SUMMARY:
The purpose of the international plastic bronchitis registry is to understand the natural course and long term health outcomes of subjects diagnosed with plastic bronchitis due to different types of casts. This provides essential data for identifying best practices and treatments. The secondary aim is to understand the structure of casts and mechanism of their formation.

DETAILED DESCRIPTION:
Plastic bronchitis (PB) patients have casts removed during bronchoscopy as part of their routine care or that they are able to expectorate (cough out) casts naturally. The casts are normally discarded. Patients that agree to participate in the registry ship the airway casts and medical history to Dr. Bruce Rubin's Research Laboratory at Virginia Commonwealth University Richmond Virginia, USA.

The lab evaluates the biopolymer composition and structure of the airway casts by immunohistochemistry in order to identify microscopic differences between expectorated casts of subjects with plastic bronchitis and sputum from other populations (cystic fibrosis,chronic obstructive pulmonary disease , and normal airways). The lab also conducts in vitro evaluation of clearability, adhesivity, cohesivity, and inflammatory mediator concentrations to better understand the nature of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Plastic bronchitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study is open to patients around the world suffering from Plastic bronchitis
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-07; Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
natural course and long term health outcomes | ongoing
  The purpose of the intrnational plastic bronchitis registry is to understand the natural course and long term health outcomes of patients diagnosed with plastic bronchitis. This provides essential data for identifying possible causes of this disease and potential treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce K Rubin, MEngr, MD, MBA, FRCPC, Principal Investigator — Children's Hospital of Richmond at VCU
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States